CLINICAL TRIAL: NCT01985490
Title: Change in Foveal Avascular Zone After Removal of Epiretinal Membrane and Internal Limiting Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-07-163
Record Dates: First submitted 2013-11-10; First posted 2013-11-15 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Epiretinal Membrane
Keywords: epiretinal membrane; foveal avascular zone; internal limiting membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- epiretinal membrane (Experimental)
  Interventions: Procedure: epiretinal membrane and internal limiting membrane removal

INTERVENTIONS:
Procedure: epiretinal membrane and internal limiting membrane removal — fluorescein angiography is performed before, 1 week, 3months and 6months after the epiretinal membrane and internal limiting membrane removal.

SUMMARY:
Fovea is characterized by its vessel-free zone, called foveal avascular zone and it can be visualized by fluorescein angiography. Removal of epiretinal membrane and internal limiting membrane is frequently performed procedure and we suspected that these procedures may affect integrity of foveal avascular zone.

The purpose of the present study is to evaluate the change of foveal avascular zone after removal of epiretinal membrane and internal limiting membrane

ELIGIBILITY:
Inclusion Criteria:

* epiretinal membrane

Exclusion Criteria:

* history of vitrectomy, intraocular surgery
* any macular disease other than epiretinal membrane
* media opacity obscuring the image of fluorescein angiography

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
area of foveal avascular zone | postoperative 6 months
  the change in area of foveal avascular zone at postoperative 6 months

SECONDARY OUTCOMES:
change in visual acuity | postoperative 6 months
change in macular thickness | at 6 months
change in metamorphopsia | postoperative 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea